CLINICAL TRIAL: NCT03344068
Title: A Single Center, Open-label, Randomized Controlled Clinical Trial on the Early and Whole Course Nutritional Support by Nutren® Optimum During Intensity Modulated Radiation Therapy for Nasopharyngeal Carcinoma
Brief Title: Early and Whole Course Nutritional Support by Nutren® Optimum During IMRT for Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Principal Investigator, Yun-fei Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-055-01
Record Dates: First submitted 2017-10-25; First posted 2017-11-17 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Nasopharyngeal Carcinoma; Nutritional Support
Keywords: nasopharyngeal carcinoma; nutritional support; early and whole course; efficacy and safety
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Intervention Model Description: The patients eligible are divided randomly. All the patients will receive radical radiotherapy with or without chemotherapy. The cases in the Experimental Group will receive Nutren® Optimum of 7 scoops tid at begin of radiotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The patients in the Experimental Group are allocated to receive radical radiotherapy with or without chemotherapy plus Nutren® Optimum of 7 scoops tid at begin of radiotherapy.
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy; Dietary Supplement: Nutren® Optimum
- Controlled Group (Active Comparator): The patients in the Controlled Group are allocated to receive radical radiotherapy with or without chemotherapy plus routine diet guidance at begin of radiotherapy.
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Intensity Modulated Radiation Therapy, Dose: GTVnx 6810cGy/30Fr, GTVnd 6400-6600cGy/30Fr, CTV1 6000cGy, CTV2 5400cGy.
Drug: Chemotherapy — Nedaplatin 80mg/m2 d1+5-fluouracil 500mg/m2 d2-5, every 3 weeks; a total of 2-3 cycles.
Dietary Supplement: Nutren® Optimum — Nutren® Optimum, 7 scoops each time, three times a day, at begin of radiotherapy
  Arms: Experimental Group

SUMMARY:
Radiation therapy remains the principal treatment for nasopharyngeal carcinoma (NPC). The most frequently occurred radiation-related side effect is probably the radiation-induced oral mucositis, which affects up to 100% of NPC patients receiving radiation therapy, especially combined with chemotherapy. Significant weight loss caused by Oral mucositis will keep patients in worse nutrition status and then to decline immune function, hematopoietic function and repair function, which will influence the patient's quality of life, reduce the tolerance of treatment, and affect treatment effect. At present, the guidelines at home and abroad more and more emphasize that early nutrition treatment and intervention before systemic malnutrition, also suggest nutrition treatment and intervention at the same time of anti-tumor treatment. First choice of nutritional intervention is oral nutrition supplement. Nutren® Optimum has a higher protein ratio and 50% of the protein sources were lactalbumin and 50% casein. Lactalbumin is a high-quality protein, with the highest nutritional value among a variety of proteins. A cup of 210ml's Nutren® Optimum contains 5g lactalbumin. Nutren® Optimum also contains dietary fiber, vitamin E, monounsaturated fat, L-carnitine, 30 kinds of vitamins and minerals and other nutrients, which can provide a comprehensive and balanced nutrition. This single center, open-label, randomized controlled clinical trial selects Nutren® Optimum as oral nutritional support for interventional group while routine diet guidance for control group, aiming to evaluate the efficacy and safety of early and whole course nutritional support by Nutren® Optimum during intensity modulated radiation therapy for nasopharyngeal carcinoma which can improve patients' nutritional state and quality of life, reduce side effects and improve the tolerability and effectiveness of antitumor treatment.

DETAILED DESCRIPTION:
Radiation therapy remains the principal treatment for nasopharyngeal carcinoma (NPC). The most frequently occurred radiation-related side effect is probably the radiation-induced oral mucositis, which affects up to 100% of NPC patients receiving radiation therapy, especially combined with chemotherapy.

Oral mucositis is just the most common cause of significant weight loss for patients with nasopharyngeal carcinoma during treatment. Patients with oral mucositis will have restriction of normal food, and alternative to semi liquid or liquid diet, resulting in inadequate nutritional intake, malnutrition, weight loss. Furthermore, worse nutrition status will decline immune function, hematopoietic function and repair function, which will influence the patient's quality of life, reduce the tolerance of treatment, and affect treatment effect.

At present, the guidelines at home and abroad more and more emphasize that early nutrition treatment and intervention before systemic malnutrition, also suggest nutrition treatment and intervention at the same time of anti-tumor treatment. Therefore, the timing of nutritional intervention changes from ineffective antitumor therapy as a palliative treatment to the early start of antitumor therapy. For nasopharyngeal carcinoma, early and whole course nutritional intervention can prevent and treat malnutrition or cachexia; improve the treatment tolerance and compliance; control or improve certain adverse reactions of radiotherapy; improve the quality of life; and then improve the function and curative effect. First choice of nutritional intervention is oral nutrition supplement. For patients without gastrointestinal dysfunction, parenteral nutrition is not necessary, even harmful, increasing the risk of infection.

Nutren® Optimum has a higher protein ratio (P:F:C = 17:35:48), and 50% of the protein sources were lactalbumin and 50% casein. Lactalbumin is a high-quality protein, which dissolved and dispersed in the whey protein. Lactalbumin is easy digestion and absorption, with high bioavailability, and net protein utilization rate (NPU) is higher than that of casein and soy protein. Lactalbumin is rich in branched chain amino acids, which can be used as energy material for energy. Lactalbumin has a sulfur-containing amino acid, which can maintain the level of GSH and be in the role of antioxidation; containing glutamine, which contributes to muscle glycogen update and improves immune function. In addition, lactalbumin can also significantly reduce neutrophil apoptosis, enhance neutrophil migration and phagocytosis, and enhance the immune function. Therefore, lactalbumin has the highest nutritional value among a variety of proteins, known as protein king. A cup of 210ml's Nutren® Optimum contains 5g lactalbumin.

Nutren® Optimum contains dietary fiber, which produces short chain fatty acids to promote the proliferation of intestinal probiotics, and play anti-inflammatory, pro-apoptotic, anti-tumor effect, and maintain intestinal health. At the same time, vitamin E is specially added in Nutren® Optimum to protect T lymphocytes, protect red blood cells, anti-oxidation, inhibit platelet aggregation, enhance immunity, and so on. In addition, 64% fat sources of Nutren® Optimum are monounsaturated fat, which conducive to the metabolism of glucose and lipid. Especially added L-carnitine can promote fat oxidation by using better fat for energy, without reducing water and muscle. Nutren® Optimum provides 30 kinds of vitamins and minerals and other nutrients, and can provide a comprehensive and balanced nutrition.

This single center, open-label, randomized controlled clinical trial selects Nutren® Optimum as oral nutritional support for interventional group while routine diet guidance for control group, aiming to evaluate the efficacy and safety of early and whole course nutritional support by Nutren® Optimum during intensity modulated radiation therapy for nasopharyngeal carcinoma, which can improve patients' nutritional state and quality of life, reduce side effects and improve the tolerability and effectiveness of antitumor treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed and previously untreated nasopharyngeal carcinoma without distant metastasis.
* Age ≥ 18 years and < 65 years.
* Karnofsky performance status (KPS) score ≥ 70.
* Planned to receive radiotherapy alone or concurrent chemoradiotherapy, with intensity-modulated radiation therapy (IMRT).
* Adequate normal organ function.
* Well nutritional status, with PG-SGA≤1 score and NRS2002<3 scores.
* Without other severe diseases.
* Signed informed consent voluntarily, and could complete required oral nutrition, questionnaire survey and follow-up.

Exclusion Criteria:

* Known allergic reaction to any component of Nutren® Optimum, or severe allergic constitution.
* Poor compliance.
* Other conditions that the investigators consider as inappropriate for enrolling into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Decline in nutritional status needed upgrading nutritional intervention | 3 months after radiotherapy
  The percentage of patients whose body weight decreased by 5% over baseline, or the PG-SGA score was more than 8, or the NRS2002 score was more than 3.

SECONDARY OUTCOMES:
Quality of life | 3 months after radiotherapy
  The standard scores assessed by EORTC QOL scale decreased by more than 10 points
Moderate and severe bone marrow depression and anemia | 3 months after radiotherapy
  Incidence of 3-4 degrees bone marrow depression and anemia according to CTCAE (version 4)
Severe oral mucositis | 3 months after radiotherapy
  Incidence of 3-4 degrees oral mucositis according to CTCAE (version 4)
Interruption rate of radiotherapy and/or chemotherapy caused by intolerance | 3 months after radiotherapy
  The percentage of patients whose radiotherapy and/or chemotherapy were interrupted by treatment-related toxicity intolerance
Complete remission | 3 months after radiotherapy
  The percentage of patients whose all the target lesions disappeared, no new lesions appeared according to RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China